CLINICAL TRIAL: NCT06827548
Title: Effect of Electrical Stimulation of the Auricular Branch of the Vagus Nerve (ABVN) on Cervical Vagus Nerve Action Potentials Phase 2 - VNS Seizure
Brief Title: ABVN Phase 2-Studying the Effect of Stimulation on the Auricular Branch of the Vagal Nerve -B
Acronym: ABVN2-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, Thomas V. Nowak, Professor of Clinical Medicine, Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006075899-B
Record Dates: First submitted 2024-12-06; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Gastro-Intestinal Disorder; Gastroparesis
MeSH Terms: conditions — Digestive System Diseases; Gastroparesis | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: vagal nerve stimulation — Cervical neck electrodes used in this part of the study will include the multi electrode array (MEA). The MEA can be placed on either side of the neck over the area of the vagus nerve to record any electrical activity that might occur during the baseline period.
  Two ECG electrodes are placed either one on each arm or on the chest for measurement of the electrocardiogram (ECG).
  Three ECG electrodes are placed on the abdomen in a line parallel to the longitudinal axis of the stomach to record the electrogastrogram (EGG).
  A onetime baseline recording will be made for 20 minutes after which the subject will be discharged from the study.
  Other Names: VNS Therapy

SUMMARY:
The purpose of this study is to find out if manual stimulation of the vagus nerve is possible. The vagus nerve is a largely-internal nerve that controls many bodily functions, including stomach function. The hope is that electrically stimulating the nerve around the external ear will also stimulate the internal vagus nerve.

DETAILED DESCRIPTION:
The purpose of this study is to find out if it is possible to gain access to the vagus nerve which is largely an internal nerve that controls stomach function. The hope is to gain access to the internal vagus nerve by electrically stimulating the nerve around the external ear. If this is possible to do this then there is hope that this will help the treatment of patients with nausea and vomiting and disordered stomach function. Healthy subjects and subjects with gastroparesis will be recruited. Subjects will undergo transcutaneous stimulation of the auricular branch of the vagus nerve and also undergo blood draw before, after stimulation and later a third draw after a period of no stimulation. Healthy subjects will also undergo vagal maneuver using the Multi Array Electrodes (MEA). Subjects will also complete health history questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with no GI symptoms
* Ages 18-80
* Undergoing VNS Therapy as part of clinical treatment for focal or partial epilepsy or seizure
* Willing to have MEA electrodes placed on the neck and bipolar electrodes placed on chest and stomach

Exclusion Criteria:

* Unable to provide consent
* Having gastric motility issues (not due to COVID 19) as determined by the PI or Sub I
* Taking medications affecting gastric motility
* Pregnant females
* Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Vagal Nerve Activation | 3 hours
  To measure the amplitude of vagal nerve compound action potentials in gastroparetic subjects with symptoms of nausea and vomiting with skin electrodes over right and left vagus nerve during ABVN stimulation and also during the vagal maneuvers phase
Measure changes in chest diameter resulting from breathing | 3 hours
  To measure and evaluate respiratory variation of heart rate.
Amplitude surface electrogastrogram | 3 hours
  To measure changes in the amplitude of the surface electrogastrogram during ABVN and also during the vagal maneuvers phase.
Heart rate variability | 3 hours
  To measure the Heart rate variability(HRV), vagal nerve compound action potentials and electrogastrogram in subjects undergoing VNS Therapy for focal or partial seizures.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas V. Nowak, MD, Principal Investigator — Professor of Clinical Medicine
Locations (1):
- Indiana University Hosptial, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT06827548/Prot_000.pdf
  • Informed Consent Form (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT06827548/ICF_001.pdf